CLINICAL TRIAL: NCT05089617
Title: To Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral Administration of YG1699 in Healthy Chinese Subjects: a Randomized, Double-blind, Placebo-controlled, Single Ascending Dose (SAD) and Multi-dose, Sequential, Bridging Study
Brief Title: To Evaluate the Safety, Tolerability, and Pharmacokinetics of YG1699（Antidiabetic） in Healthy Chinese Sbjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Youngene Therapeutics Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: YG1699-102
Record Dates: First submitted 2021-09-26; First posted 2021-10-22 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Single Ascending Dose and Multiple Dose
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAD Cohort 1 (Experimental): 5 mg YG1699 or Placebo
  Interventions: Drug: YG1699
- SAD Cohort 2 (Experimental): 25 mg YG1699 or Placebo
  Interventions: Drug: YG1699
- Multiple Doses Cohort 1 (Experimental): 20 mg YG1699 or Placebo
  Interventions: Drug: YG1699

INTERVENTIONS:
Drug: YG1699 — YG1699 is a novel investigational dual inhibitor of sodium-dependent glucose cotransporters, SGLT1 and SGLT2, indicated as an adjunct to diet and exercise to improve glycemic control and weight loss in adults with T2DM. A subsequent indication will be developed for YG1699 to improve glycemic control in adults with T1DM.
  Drug: Placebo
  Placebo is the same appearance as YG1699.

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multi-dose, sequential, bridging study in healthy volunteer using YG1699 .

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dose-ascending study to evaluate the safety, tolerability, and pharmacokinetics (PK) of YG1699 following single ascending and multiple oral dose administration.

The study consists of 2 parts: Part 1, SAD dose- ascending; Part 2, multi-dose ascending.

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of giving informed consent and complying with study procedures;
2. Are between the ages of 18 and 55 years, inclusive;
3. Female subjects have a negative urine pregnancy test result at screening and Day 0, and meet one of the following criteria:

   1. Using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives) [e.g., hormonal contraceptives (oral, patch, injectable or vaginal ring), implantable device (implantable rod or intrauterine device), or a double barrier (e.g., diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge)]
   2. Surgically sterile for at least 3 months prior to screening by one of the following means:

      Bilateral tubal ligation Bilateral salpingectomy (with or without oophorectomy) Surgical hysterectomy Bilateral oophorectomy (with or without hysterectomy)
   3. Postmenopausal, defined as the following:

   Last menstrual period greater than 12 months prior to screening Postmenopausal status confirmed by serum Follicle-Stimulating Hormone（FSH） and estradiol levels at screening;
4. Considered healthy by the Investigator, based on subject's reported medical history, full physical examination, clinical laboratory tests, 12-lead ECG, and vital signs;
5. Non-smoker and less than 5 cigarettes/day or nicotine replacement products in last 6 months;
6. Body mass index (BMI) of 18.0 to 30.0 kg/m2 inclusive and body weight not less than 50 kg;
7. Male subjects with female partners of child bearing potential must agree to use condoms for the duration of the study and until 12 weeks after dosing with the study drug and must refrain from donating sperm for this same period.

Exclusion Criteria:

1. Subjects of non-Chinese nationality living or working in China, or persons of non-East Asian descent who are Chinese nationals;
2. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator;
3. History of food or drug allergy;
4. Known or suspected malignancy;
5. History of unexplained syncope, symptomatic hypotension or hypoglycemia;
6. History or family history of long corrective QT interval（QTc） syndrome;
7. History of chronic diarrhea, malabsorption, unexplained weight loss, food allergies or intolerance;
8. Poor venous access;
9. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C antibody or treponema pallidum antibody ;
10. Donated or lost >500ml of blood in the previous 3 months;
11. Taken an investigational drug or participated in a clinical trial within 3 months (or 5 half-lives), whichever is longer;
12. Taken any prescription medications within 14 days or 5 half-lives (whichever is longer) of the first dose of study drug;
13. Hospital admission or major surgery within 6 months prior to screening;
14. A history of prescription drug abuse within 9 months prior to screening;
15. A history of alcohol abuse according to medical history within 9 months prior to screening;
16. Female subjects with positive pregnancy test, pregnant or breastfeeding;
17. A positive screen for alcohol, drugs of abuse at screening;
18. An unwillingness or inability to comply with food and beverage restrictions during study participation;
19. Use of over-the-counter (OTC) medication and herbal within 7 days prior to dosing (Note: Use of acetaminophen at < 2 g/day is permitted until 24 hours prior to dosing);
20. Any condition or finding that in the Investigators opinion would put the subject or study conduct at risk if the subject were to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-01-09 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Adverse events will be evaluated | 81 Days
  Safety and Tolerability of YG1699

SECONDARY OUTCOMES:
Area Under the Curve [AUC] | 81 Days
  area under the plasma drug concentration time curve from time 0 to T (AUC)
maximum plasma concentration (Cmax) | 81 Days
  maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jiaojuan He, Master, Study Director — Youngene Therapeutics Inc., Ltd.
Locations (1):
- Shanghai Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No